CLINICAL TRIAL: NCT02918253
Title: HDR Monotherapy for Prostate Cancer: A Feasibility Study of Focal Radiotherapy Yields
Brief Title: HDR Focal: Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-5490
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: High dose-rate brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tumour visible on MRI (Experimental): Targeted focal HDR Brachytherapy to dominant lesion +/- whole-gland elective dose
  Interventions: Radiation: targeted focal HDR brachytherapy
- No tumour visible on MRI (Active Comparator): Whole-gland HDR Brachytherapy
  Interventions: Radiation: Whole-gland HDR Brachytherapy

INTERVENTIONS:
Radiation: targeted focal HDR brachytherapy
  Arms: Tumour visible on MRI
Radiation: Whole-gland HDR Brachytherapy — Control/Standard of Care
  Arms: No tumour visible on MRI

SUMMARY:
Brachytherapy as a monotherapy treatment is highly effective for localized prostate cancer, traditionally being delivered to the whole prostate gland. Lately, low dose rate (LDR) brachytherapy has been increasingly replaced by high dose rate (HDR) brachytherapy treatment schemes. While brachytherapy's oncologic outcomes are excellent, it is not without incidence adverse effects including urinary, rectal, and sexual toxicities that affect the patient's quality of life.

This study will incorporate HDR monotherapy treatment option for early stages and favourable risk prostate cancer.

Additionally, we aim to evaluate the role of focal HDR brachytherapy for well-defined disease based on multiparametric MRI (mpMRI). This approach may offer an option of reducing the treatment toxicities while maintaining oncologic outcomes when compared with whole-gland therapy. Advantages in quality of life could be exhibited in the form of reduced urinary discomfort and incontinence, rectal symptoms, and improved erectile and prostatic gland function. This study would be particularly relevant in the current era of earlier localized prostate cancer detection, where newer imaging modalities (e.g. mpMRI) become a routine component of patient care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ECOG performance status 0 - 2
* Histological evidence of prostate adenocarcinoma
* Low- and favorable intermediate-risk prostate cancer
* Informed consent: All patients must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed
* No contraindications to MRI:
* Absent or unifocal intraprostatic disease (<2 separate/distinct lesions), on multiparametric MRI
* Prostate gland size <80cc
* Baseline IPSS <18
* No TRUP within the past 6 months, nor large TURP defect
* Absence of radiological evidence of regional or distant metastases (optional evaluation, at physician discretion)
* No previous pelvic and/or prostate EBRT and/or brachytherapy
* No contraindications to general anesthesia, or spinal/epidural anesthesia
* Absence of bleeding diathesis and/or anti-coagulative therapy that cannot be temporarily ceased during brachytherapy
* No contraindications to endorectal coil, surgically absent rectum, severe hemorrhoids or colorectal surgery
* Negative past medical history of Ulcerative Colitis, Crohn's Disease, Ataxia Telangiectasia, or SLE
* Absence of latex allergy
* No other medical conditions deemed by the PI to make patient ineligible for prostate HDR brachytherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10-14 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
number of patients achieving biochemical control | 2 yrs

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No